CLINICAL TRIAL: NCT05311475
Title: A Multicenter, Randomized, Double-blind, Placebo and Active Controlled Parallel-group Trial to Assess the Efficacy and Safety of the Fixed Combination Medicinal Product Mometasone Furoate + Azelastine Hydrochloride Nasal Spray (50 + 140 mcg) in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Prospective, Randomized, Multinational, Multicenter, Double-blind, Placebo and Active Controlled Trial in 4 Parallel-groups of Patients Suffering From Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLK21001/SAN-0677; 2021-004050-31 (EudraCT Number)
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate; azelastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mometasone + Azelastine (Experimental): Mometasone + Azelastine (50 + 140 mcg per actuation)
  Interventions: Drug: Mometasone; Drug: Azelastine
- Mometasone (Active Comparator): Mometasone furoate nasal spray (50 mcg per actuation)
  Interventions: Drug: Mometasone
- Azelastine (Active Comparator): Azelastine hydrochloride nasal spray (140 mcg per actuation)
  Interventions: Drug: Azelastine
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone — Mometasone furoate nasal spray (50 mcg per actuation)
  Arms: Mometasone; Mometasone + Azelastine
Drug: Azelastine — Azelastine hydrochloride nasal spray (140 mcg per actuation)
  Arms: Azelastine; Mometasone + Azelastine
Drug: Placebo — Placebo nasal spray
  Arms: Placebo

SUMMARY:
The trial will be conducted as a prospective, randomized, multinational, multicenter, double-blind, placebo and active controlled trial in 4 parallel-groups of patients suffering from seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

Only patients fulfilling all of the following criteria at screening Visit 1 should be included in the present trial:

* Male or non-pregnant, non-lactating female patient aged between 12 and 65 years (valid for Poland) OR between 18 and 65 years (valid for Bulgaria, Moldova and Germany) inclusive on the date of consent.
* Female patient of childbearing potential abstaining from sexual intercourse or using a reliable method of contraception (e.g., condom with spermicide, intra uterine device, oral, injected, transdermal or implanted hormonal contraceptives, or had in the past a female sterilization e.g. tubal ligation, hysterectomy, oophorectomy, salpingectomy) for 30 days before enrolment and agree to continue its use during the trial.
* A minimum of two seasons of previous history of at least moderate seasonal allergic rhinitis (SAR) to the pollen/allergens in season at the time the trial is being conducted.
* Patient must have the following SAR symptoms: (i) nasal congestion, and at least one of the following; (ii) rhinorrhea; (iii) nasal itching; or (iv) sneezing. Nasal congestion plus one other nasal symptom score both rated by the patient as at least moderate in severity (≥2 on a 0-3 scale) and Total Nasal Symptom Score (TNSS) ≥6.0 over the last 24 hours.
* Negative SARS-CoV-2 Rapid Antigen Test result at screening visit.
* For adults (≥18 years): Informed consent to participate in the trial provided in written form; For adolescents (≥12 - <18 years): own patient informed consent/ assent to participate in the trial and the informed consent from all parent(s)/ legal guardian(s) provided in written form.

Inclusion criteria at Visit 2 (selection for randomization):

Only patients fulfilling at Visit 2 the following inclusion criteria will be randomized in the trial:

* Pollen-specific immunoglobulin E (sIgE) test ≥EAST class 3 (at least 3.5 kU/l).
* Negative serum (hCG) pregnancy test (for female patient only).
* Patient selected for randomization must have the following SAR symptoms over 3 days during the 3- to 5-day baseline period: (i) nasal congestion, and 1 or more of the following; (ii) rhinorrhea; (iii) nasal itching; or (iv) sneezing.
* The mean TNSS must be ≥6.0 over 3 days out of the last 3-5 days of the Placebo run-in period; additionally, the mean nasal congestion score and mean of 1 other nasal symptom score both must be ≥2 (on a 0-3 scale) over 3 days out of the last 3-5 days of the Placebo run-in period.

Exclusion Criteria:

Patients presenting any of the following criteria will NOT be included in the trial:

* Simultaneous participation in other clinical trials.
* Use of any investigational drug within 30 days prior to enrolment (Visit 1).
* Clinically significant medical condition (such as cardiovascular, hepatic, neurological, hematological, renal, gastrointestinal, endocrine or other major systemic disease) that, in the judgement of the investigator, would interfere with the trial, require treatment, or make implementation of the protocol or interpretation of the trial results difficult.
* Any known hypersensitivity to azelastine or other antihistamines, mometasone or other steroids, or any of the components of the trial nasal sprays.
* Structural nasal abnormalities symptomatic enough to cause nasal obstruction, as judged by the investigator, or any recent nasal surgery or trauma that is not completely healed.
* Any other nasal conditions, including infectious rhinitis, sinusitis, rhinitis medicamentosa, atrophic rhinitis, and perennial rhinitis (PAR) (coexisting PAR will be allowed if SAR shows clear exacerbations).
* History of upper respiratory tract or sinus infection that required antibiotic therapy with the last dose within 14 days prior to screening.
* Treatment for oral candidiasis within 30 days of starting the trial.
* Presence of untreated fungal, bacterial or viral systemic infection, or infection of the ear, nose, and throat or oral cavity of any character.
* Presence of ocular herpes simplex or cataracts, or a history of glaucoma.
* Vaccination within 14 days prior to screening visit.
* History of habitual abuse of nasal decongestants (rhinitis medicamentosa).
* History of non-response to intranasal steroids.
* History of non-response to antihistamines.
* Recent exposure or being at risk to chicken pox or measles exposure.
* The patient is receiving immunotherapy or has received immunotherapy in the last 24 months.
* Use of anti-immunoglobulin E antibodies within 6 months prior to screening visit.
* Use of any of the following drugs:

  1. Systemic corticosteroid therapy within 60 days prior to screening visit.
  2. Topical (intranasal, inhaled, ocular) corticosteroid therapy within 30 days prior to screening visit.
  3. Immunosuppressive drugs and immunomodulating drugs (e.g., omalizumab, mepolizumab or dupilumab) within 30 days prior to screening visit.
  4. Cromolyn sodium or nedocromil within 14 days prior to screening visit.
  5. Tricyclic antidepressants within 14 days prior to screening visit.
  6. Histamine H1 antagonists (any generation of antihistamines) i.e., loratadine, cetirizine, desloratadine, levocetirizine, fexofenadine, hydroxyzine, etc. within 14 days prior to screening visit.
  7. Leukotriene modifiers within 7 days prior to screening visit.
  8. Nasal or oral decongestants (including anticholinergic agents, oxymetazoline, ephedrine or pseudoephedrine, and other vasoconstrictors) and mucolytics (like guaifenesin), or other medications that could mask the symptoms of rhinitis, e.g., major tranquilizers, anti-epileptic agents, within 3 days prior to screening visit. This includes over-the-counter preparations for common cold or eye drops containing any of the above-mentioned agents.
  9. Nasal sprays or washes with any medication, including saline, within 24 hours prior to screening visit.
* Planned to travel outside of the geographical region (as judged by the investigator according to regional pollination calendar) for >3 consecutive days during the trial.
* Member of the investigational trial staff or a member of the family of the investigational trial staff.
* History of alcohol or drug abuse within the last 5 years.
* History of non-compliance with medication regimens or treatment protocols in previous clinical studies.
* Legal incapacity (for adults only) and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequences of the trial.
* Patients who are known or suspected to be in custody or submitted to an institution due to a judicial order.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the daily Total Nasal Symptom Score (TNSS) | Baseline, Day 7
  The benefit of the treatment with the fixed combination medicinal product Momeatsone+Azelastine nasal spray (test product) in comparison to the treatment with the individual medicinal products Mometasone nasal spray and Azelastine nasal spray (comparator products) will be assessed by comparing the change from baseline in the daily Total Nasal Symptom Score (TNSS) during the first seven days of treatment. Total Nasal Symptom Score (TNSS) of 4 symptoms (rhinorrhea, sneezing, nasal itching, and nasal congestion) will be assessed by the patient in a patient's diary. Each symptom will be scored on a 4-point scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms, such that the maximum TNSS is 12.

SECONDARY OUTCOMES:
Change from baseline in the daily Total Nasal Symptom Score (TNSS) | Baseline, Day 14
  Total Nasal Symptom Score (TNSS) of 4 symptoms (rhinorrhea, sneezing, nasal itching, and nasal congestion) will be assessed by the patient in a patient's diary starting at Visit 1 for the baseline run-in period (3 to 5 days). The mean of the symptom scores during the last 3 days prior to Visit 2 will be used to calculate baseline symptoms. Following randomization at Visit 2, the patient will document the TNSS in the evening retrospectively for each day of treatment until treatment day 14. Each symptom will be scored on a 4-point scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms, such that the maximum TNSS is 12.
Change from baseline in individual daily nasal symptoms | Baseline, Day 7 and Day 14
  Change from baseline in individual daily nasal symptoms (nasal congestion, rhinorrhea, nasal itching and sneezing) during 7 and 14 days of treatment for all four arms will be assessed.
Change from baseline in individual daily ocular symptoms | Baseline, Day 7 and Day 14
  Ocular itching and Redness and Ocular tearing will be scored on a 4-point scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The symptoms will be assessed by the patient in a patient's diary starting at Visit 1. The patient will document the ocular symptoms in the evening retrospectively for each day of treatment until treatment day 14.
Baseline-adjusted differences in nasal obstruction assessed by peak nasal inspiratory flow measurements (PNIF) | Baseline, Day 7 and Day 14
  The PNIF will be performed by means of portable In-Check Nasal flow meter using a face mask which the patient applies over the nose (without touching it) with the mouth closed. The In-Check Nasal is a portable inspiratory flow meter, measuring inspiratory flow between 30-370 L/min.
Change from baseline in Rhinoscopy score | Baseline, Day 7 and Day 14
  Rhinoscopy score: during the nasal examination the investigator will evaluate the symptoms rhinorrhea, redness and edema using a 4-point scale as follows: absent = 0, mild = 1, moderate = 2, and severe = 3.
Intra-group changes in health-related Quality of Life (RQLQ) | Baseline, Day 7 and Day 14
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) has 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). There are 3 'patient-specific' questions in the activity domain which allow patients to select 3 activities in which they are most limited by their rhinoconjunctivitis. Patients recall how bothered they have been by their rhinoconjunctivitis during the previous week and to respond to each question on a 7-point scale (0 = not impaired at all - 6 = severely impaired). The overall RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains.
Number of responders with an improvement of ≥ 0.5 points in the assessment of overall RQLQ | Baseline, Day 7 and Day 14
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) has 28 questions in 7 domains (activity limitation, sleep problems, nose symptoms, eye symptoms, non-nose/eye symptoms, practical problems and emotional function). There are 3 'patient-specific' questions in the activity domain which allow patients to select 3 activities in which they are most limited by their rhinoconjunctivitis. Patients recall how bothered they have been by their rhinoconjunctivitis during the previous week and to respond to each question on a 7-point scale (0 = not impaired at all - 6 = severely impaired). The overall RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains.
Intra-group changes in the Rhinitis Control Assessment Test (RCAT) score | Baseline, Day 7 and Day 14
  Rhinitis Control Assessment Test (RCAT) questionnaire has 6 items that include nasal congestion, sneezing, watery eyes, sleep problems caused by rhinitis, activity avoidance, and nasal or other allergy symptoms control. Responses are measured on a 5-point scales. RCAT scores range from 6 to 30, with higher scores indicating better rhinitis control.
Number of responders with a RCAT score ≥22 | Baseline, Day 7 and Day 14
  Rhinitis Control Assessment Test (RCAT) questionnaire has 6 items that include nasal congestion, sneezing, watery eyes, sleep problems caused by rhinitis, activity avoidance, and nasal or other allergy symptoms control. Responses are measured on a 5-point scales. RCAT scores range from 6 to 30, with higher scores indicating better rhinitis control.
Onset of action: Instantaneous TNSS | On Day 2 (first day of treatment) from 0 to 8 hours (at 5 minutes, 15 minutes, 30 minutes, 1 h, 2 h, 4 h, 8 h) after the first dose administration
  Instantaneous Total Nasal Symptom Score (TNSS) of 4 symptoms (rhinorrhea, sneezing, nasal itching, and nasal congestion) will be assessed by the patient in a patient's diary.
Onset of action: instantaneous ocular symptoms | On Day 2 (first day of treatment) from 0 to 8 hours (at 5 minutes, 15 minutes, 30 minutes, 1 h, 2 h, 4 h, 8 h) after the first dose administration
  Instantaneous Ocular itching and Redness and Ocular tearing will be scored on a 4-point scale where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (27):
- Bulgaria (6):
  - Sandoz Investigative Site, Burgas
  - Sandoz Investigative Site, Gabrovo
  - Sandoz Investigative Site, Plovdiv
  - Sandoz Investigative Site, Sliven
  - Sandoz Investigative Site, Sofia
  - Sandoz Investigative Site, Varna
- Germany (10):
  - Sandoz Investigative Site, Aachen
  - Sandoz Investigative Site, Dreieich
  - Sandoz Investigative Site, Dresden
  - Sandoz Investigative Site, Duisburg
  - Sandoz Investigative Site, Hamburg
  - Sandoz Investigative Site, Heidelberg
  - Sandoz Investigative Site, Neuenhagen
  - Sandoz Investigative Site, Röthenbach
  - Sandoz Investigative Site, Schorndorf
  - Sandoz Investigative Site, Viernheim
- Sandoz Investigative Site, Chisinau, Moldova
- Poland (10):
  - Sandoz Investigative Site, Brzeg Dolny
  - Sandoz Investigative Site, Chodzież
  - Sandoz Investigative Site, Inowrocław
  - Sandoz Investigative Site, Jaksice
  - Sandoz Investigative Site, Lodz
  - Sandoz Investigative Site, Lublin
  - Sandoz Investigative Site, Ostrowiec
  - Sandoz Investigative Site, Poznan
  - Sandoz Investigative Site, Warsaw
  - Sandoz Investigative Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com